CLINICAL TRIAL: NCT05445817
Title: Pulmonary Care and Research Collaborative Patient Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pulmonary Care and Research Collaborative Limited (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ILDC-001
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Interstitial Lung Disease
Keywords: Progressive Fibrosing Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis; Interstitial Lung Disease Associated With Systemic Sclerosis; Myositis-Associated Interstitial Lung Disease; Sarcoidosis; Hypersensitivity Pneumonitis; Pulmonary Fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis; Sarcoidosis; Alveolitis, Extrinsic Allergic; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research study is to build and maintain a registry of people with interstitial lung disease (ILD). Medical information collected for this registry may be used to advance ILD and pulmonary research and improve patient care. This is an observational registry. Participants will not receive any investigational treatments or investigational drugs as part of their participation in this registry.

DETAILED DESCRIPTION:
The registry will contain longitudinal medical histories of ILD patients. The creation and curation of the registry with utilize release of information services, biomedical informatics methods and human expert reviews. Among the registry's long-term goals is to utilize its data and informatics resources to study and advance ILD diagnosis and treatment. The registry will be developed with a set of capabilities to consistently, repeatedly, and economically build research-grade datasets that allow cohort development from natively unstructured and non-standard phenotypic clinical and imaging data.

ELIGIBILITY:
Inclusion Criteria:

* People with a confirmed diagnosis of interstitial lung disease by a primary care physician and/or pulmonologist.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with a confirmed diagnosis of interstitial lung disease by a primary care physician and/or pulmonologist.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Development and implementation of a database populated with de-identified longitudinal medical histories of interstitial lung disease patients. | Up to 18 months

SECONDARY OUTCOMES:
Advancing the understanding of the natural course and the treatments of interstitial lung diseases. | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Barakat, PhD, Principal Investigator — Pulmonary Care and Research Collaborative, Ltd.
Locations (1):
- Pulmonary Care and Research Collaborative, Ltd., Boston, Massachusetts, United States